CLINICAL TRIAL: NCT02596022
Title: The Effect of Glutamatergic Modulation on Cocaine Self-administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Elias Dakwar, research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6716
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CI-581a (Experimental): Administration of CI-581a followed 2 weeks later by CI-581b
  Interventions: Drug: CI-581a; Drug: CI-581b
- CI-581b (Active Comparator): Administration of CI-581b followed 2 weeks later by CI-581a
  Interventions: Drug: CI-581a; Drug: CI-581b

INTERVENTIONS:
Drug: CI-581a — a 50 minute infusion 24 hours prior to cocaine self-administration session
Drug: CI-581b — a 50 minute infusion 24 hours prior to cocaine self-administration session

SUMMARY:
Repeated drug consumption may progress to problematic use by triggering neuroplastic adaptations that attenuate sensitivity to natural rewards while increasing reactivity to craving and drug cues. Converging evidence suggests that glutamate modulation may work to correct these adaptations and rapidly restore motivation for delayed non-drug rewards relative to immediate drug use. Using an established laboratory model aimed at evaluating behavioral shifts in the salience of cocaine now vs. money later, the investigators will test the effect of CI-581a on cocaine self-administration as compared to the active control.

ELIGIBILITY:
Inclusion Criteria:

1. Active cocaine dependence with at least 8 days of use or at least 4 binges of large amounts (>$200/occasion) over the past 30 days, and displaying at least one positive utox during screening
2. Physically healthy
3. No adverse reactions to study medications
4. 21-55 years of age
5. Capacity to consent and comply with study procedures, including sufficient proficiency in English
6. Not seeking treatment

Exclusion Criteria:

1. Meets DSM IV criteria for current major depression, bipolar disorder, schizophrenia, any psychotic illness, including substance induced psychosis, and current substance-induced mood disorder with HAMD score > 12.
2. Physiological dependence on another substance, such as alcohol, opioids, or benzodiazepines, excluding caffeine, nicotine, and cannabis
3. Delirium, Dementia, Amnesia, Cognitive Disorders, or Dissociative disorders
4. Current suicide risk or a history of suicide attempt within the past year
5. Pregnant or interested in becoming pregnant during the study period
6. Any of the following cardiac conditions: clinically significant left ventricular hypertrophy, angina, clinically significant arrhythmia, or mitral valve prolapse
7. Unstable physical disorders which might make participation hazardous such as end-stage AIDS, hypertension (>140/90), WBC < 3.5, active hepatitis or other liver disease with elevated transaminase levels (< 2-3 X upper limit of normal will be considered acceptable if PT/PTT is normal), renal failure (creat > 2, BUN >40), or untreated diabetes
8. Previous history of ketamine or midazolam misuse or abuse, and a history of an adverse reaction/experience with prior exposure to cocaine, ketamine or midazolam
9. Recent history of significant violence (past 2 years)
10. Abnormal pseudocholinesterase level
11. First degree relative with a psychotic disorder (bipolar disorder, schizophrenia, schizoaffective disorder, or psychosis NOS)
12. BMI > 35, or a history of documented obstructive sleep apnea
13. On psychotropic or other medications whose effect could be disrupted by participation in the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — Columbia College of Physicians and Surgeons

RESULTS

PARTICIPANT FLOW:
Groups:
- CI-581a First, Followed by CI-581b: Administration of CI-581a followed 2 weeks later by CI-581b
  CI-581a: a 50 minute infusion 24 hours prior to cocaine self-administration session
  CI-581b: a 50 minute infusion 24 hours prior to cocaine self-administration session
- CI-581b First, Followed by CI-581a: Administration of CI-581b followed 2 weeks later by CI-581a
  CI-581a: a 50 minute infusion 24 hours prior to cocaine self-administration session
  CI-581b: a 50 minute infusion 24 hours prior to cocaine self-administration session
Period: Overall Study
Arm/Group | CI-581a First, Followed by CI-581b | CI-581b First, Followed by CI-581a
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CI-581a First, Followed by CI-581b | CI-581b First, Followed by CI-581a | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (6.1) | 48.6 (6.1) | 48.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Choices to Self-administer Cocaine (Out of 5 Choices)
Description: Participants provided 5 choices (cocaine 25 mg now vs. $11 later), with choices spaces 15 minutes apart over the course of the session.
Time Frame: 24 hours post-infusion
Measure: Mean (Standard Deviation); unit: number of cocaine choices
Arm/Group | CI-581a | CI-581b
Number analyzed (Participants) | 18 | 18
number of cocaine choices | 1.61 (1.3) | 4.33 (1.8)

ADVERSE EVENTS:
Time Frame: 6 weeks.
Arm/Group | CI-581a First, Followed by CI-581b | CI-581b First, Followed by CI-581a
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No